CLINICAL TRIAL: NCT06598683
Title: Effects Of Transcranial Direct Current Stimulation On Spasticity In Stroke Patients
Brief Title: tDCS and Spasticity in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC02039 Aqsa Liaqat
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; spasticity; transcranial direct current stimulation
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Transcranial Direct Current Stimulation; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental)
  Interventions: Other: tDCS; Other: Conventional
- Conventional (Active Comparator)
  Interventions: Other: Conventional

INTERVENTIONS:
Other: tDCS — Stimulation in each session will be applied for 20 min by two 5 × 4 cm (20 cm2) saline-soaked sponge electrodes at an intensity of 1.5 mA (0.075 mA/cm2). A gradual ramp up and down of stimulation for 10 s at the beginning and the end of stimulation
  Arms: tDCS
Other: Conventional — ROM exercises for upper and lower extremities, Stretching of agonists, Strengthening of antagonists, Core stability exercises, Static and dynamic balance activities, Gait training, Functional training

SUMMARY:
Multiple research has worked on tDCS and its impact on stroke. But none have studied the effects of tDCS on stroke in relation to the different stages of stroke like mild, moderate, moderate to severe and severe stroke as per national institute of health (NIH) scale.

Additionally, this study will be conducted to address the few drawbacks in previous studies such as short follow up period by employing evidence based standardized protocols. It can potentially instigate the efficacy of tDCS on spasticity, motor recovery and Quality of life in relation to the different severity levels of stroke.

DETAILED DESCRIPTION:
Multiple noninvasive brain stimulation is also introduced over the few years regarding their impact on spasticity, tDCS being the most common due to its effects on spasticity. There are multiple structural and functional changes in motor cortex post stroke, tDCS causes improvement in motor control by reorganizing the motor cortex. Anodal and cathodal tDCS are based on the current direction with cathodal decreasing excitability of the cortex area and anodal increasing it. Anodal tDCS is more effective in reducing spasticity as compared to cathodal. The change in cortical excitation alters the reflex arc i.e. altering the neurons and reducing their excitability which causes a decrease in tone and facilitates neuroplasticity.

Spasticity is often found along with weakness in stroke and is one of the reasons for impaired motor function, increased resistance to stretch and is due to increased excitability and abnormal regulation of spindle and reflex arc. With chronicity and reduced motor control spasticity also increases by 97 %. Spasticity and paresis lead to impaired motor control. Spasticity will not change recovery in function in early stages but is going to affect motor recovery in all stages. Spasticity disrupts motor function and the daily tasks which creates different levels of dependence in the patients hence effecting the QOL. Spasticity is found in almost 40% of individuals suffering from stroke. It affects joints and extremities in a way that impedes function and ADLs. Painful, restricted joints resulting from prolonged spasticity badly impacts the QOL leading to high burden on caregivers

ELIGIBILITY:
Inclusion Criteria:

* Stroke for more than 6 months.
* Both genders.
* Spasticity score ≥1 at modified ashworth scale.
* National Institutes of Health Stroke Scale (NIHSS) for severity level; Mild (1-4), Moderate (5-15), Moderate to Severe (16-20), Severe (21-42)

Exclusion Criteria:

* Have any metallic implant including intracranial electrode, pacemaker, surgical clip.
* Any symptoms effecting understanding of instructions.
* Any neurological disorder

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 8 week
  MAS is a tool to measure hypertonia. It scores the resistance on a 5 point ordinal scale with an increase value indicating hypertonia. Intrarater reliability of MAS was found to be good to excellent for upper (k= 0.71-0.94) and lower extremities(k= 0.55-0.97) while interrater reliability was poor to moderate for upper (k= 0.25-0.66)and lower extremities (k= 0.41-0.54)
Fugl Meyr Assessment | 8 week
  FMA is used for the assessment of physical performance and sensorimotor function of neurological patients. It uses a 3-point ordinal scale to score individuals' ability to perform a certain task. Total score is 226. It has excellent inter and intrarater reliability. (ICC 0.95)

SECONDARY OUTCOMES:
SS-QoL | 8 week
  It is used for estimating the quality of life of stroke patients. It contains 49 questions related to different personal and social aspects. Scoring is done on a ordinal scale of 1-5 with an increase score indicating independence. It is a valid and reliable tool to use in stroke population (Cronbach's alpha 0.903)

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Pakistan Railway General Hospital, Rawalpindi, Punjab Province
  - Pakistan Railway Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng H, Chen J, Guo Y, Tan S. Prevalence and Risk Factors for Spasticity After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Jan 20;11:616097. doi: 10.3389/fneur.2020.616097. eCollection 2020. PMID 33551975
- [Background] Cheng H, Fang X, Liao L, Tao Y, Gao C. Prevalence and factors influencing the occurrence of spasticity in stroke patients: a retrospective study. Neurol Res. 2023 Feb;45(2):166-172. doi: 10.1080/01616412.2022.2127249. Epub 2022 Sep 25. PMID 36153827
- [Background] Lackritz H, Parmet Y, Frenkel-Toledo S, Banina MC, Soroker N, Solomon JM, Liebermann DG, Levin MF, Berman S. Effect of post-stroke spasticity on voluntary movement of the upper limb. J Neuroeng Rehabil. 2021 May 13;18(1):81. doi: 10.1186/s12984-021-00876-6. PMID 33985543
- [Background] Li S, Francisco GE, Rymer WZ. A New Definition of Poststroke Spasticity and the Interference of Spasticity With Motor Recovery From Acute to Chronic Stages. Neurorehabil Neural Repair. 2021 Jul;35(7):601-610. doi: 10.1177/15459683211011214. Epub 2021 May 12. PMID 33978513
- [Background] Wang X, Ge L, Hu H, Yan L, Li L. Effects of Non-Invasive Brain Stimulation on Post-Stroke Spasticity: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Brain Sci. 2022 Jun 27;12(7):836. doi: 10.3390/brainsci12070836. PMID 35884643